CLINICAL TRIAL: NCT01650857
Title: Pulmonary Hypertension: Efficacy of a 3 Week Inpatient Pulmonary Rehabilitation on Physical Condition, Body Composition and Health Related Quality of Life - an Observational Study
Brief Title: Pulmonary Hypertension: Efficacy of a 3 Week Inpatient Rehabilitation on Physical Condition, Body Composition and Health Related Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hannover Medical School (Other)
Collaborators: Klinik Bad Fallingbostel (Unknown)
Responsible Party: Principal Investigator, Martin G Dierich, MD, MD, Hannover Medical School
Other Study IDs: HannoverMS PH-Reha001
Record Dates: First submitted 2012-07-21; First posted 2012-07-26 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Pulmonary Hypertension: Efficacy of Rehabilitation
Keywords: Pulmonary hypertension; Rehabilitation; Exercise capacity; Body composition; Health related Quality of Life
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pulmonary hypertension (PH) leads to impaired physical condition (PC), body composition (BC) and health-related quality of life (HRQOL). We hypothesized that a 3 week inpatient pulmonary rehabilitation (PR) improves PC, BC and HRQOL.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) impairs physical condition (PC), body composition (BC) and health-related quality of life (HRQOL).

Specific pharmacological treatment and - in selected patients, refractory to agents - lung or combined heart and lung transplantation can improve physical functioning and long term survival. Initial trials with limited numbers of patients were encouraging. Investigation of larger cohorts is essential to assess the efficacy of rehabilitation programmes in PH.

We hypothesize that a 3 week inpatient pulmonary rehabilitation (PR) improves PC, BC and HRQOL in patients with PH in functional classes (FC) II and III. Critical ill patients with a functional class IV are excluded. All patients with PH undergo a 3-week inpatient rehabilitation program (interval bicycle and strength training, physiotherapy, psychological support, education). Exercise testing (peak work load (PWL) 6-min-walk distance), body composition (bioimpedance analysis BIA: lean body mass (LBM), body cell mass (BCM), BCM/LBM ratio, phase angle (PA)) and HRQOL (SF 36 questionnaire) are assessed at baseline and completion of PR.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pulmonary hypertension
* Functional class II-III

Exclusion Criteria:

* Functional class I and IV
* Right heart decompensation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary hypertension in World Heart Organization functional classification classes (FC) II and III
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | 3 weeks
  Exercise capacity (peak work load and 6-minute walk distance at completion of an 3-week inpatient pulmonary rehabilitation)

SECONDARY OUTCOMES:
Body composition | 3 weeks
  Body composition (bioimpedance analysis)

OTHER OUTCOMES:
Health related Quality of Life | 3 weeks
  Health related Quality of Life (Short form 36 questionnaire)
Right ventricular function | 3 weeks
  Right ventricular function (echocardiography: estimated right ventricular systolic pressure, Tricuspid annular plane systolic excursion, left ventricular eccentricity index)
Activities of daily living | 3 weeks
  Activities of daily living (Barthel's Index)

CONTACTS AND LOCATIONS:
Overall Officials: Martin G Dierich, MD, Principal Investigator — Department of Respiratory Diseases, Hannover Medical School
Locations (1):
- Klinik Bad Fallingbostel, Bad Fallingbostel, Lower Saxony, Germany

REFERENCES:
- [Background] Rosenkranz S, Ghofrani HA, Grunig E, Hoeper MM. Cologne Consensus Conference on pulmonary hypertension. Int J Cardiol. 2011 Dec;154 Suppl 1:S1-2. doi: 10.1016/S0167-5273(11)70487-9. No abstract available. PMID 22221968
- [Background] Task Force for Diagnosis and Treatment of Pulmonary Hypertension of European Society of Cardiology (ESC); European Respiratory Society (ERS); International Society of Heart and Lung Transplantation (ISHLT); Galie N, Hoeper MM, Humbert M, Torbicki A, Vachiery JL, Barbera JA, Beghetti M, Corris P, Gaine S, Gibbs JS, Gomez-Sanchez MA, Jondeau G, Klepetko W, Opitz C, Peacock A, Rubin L, Zellweger M, Simonneau G. Guidelines for the diagnosis and treatment of pulmonary hypertension. Eur Respir J. 2009 Dec;34(6):1219-63. doi: 10.1183/09031936.00139009. Epub 2009 Sep 12. No abstract available. PMID 19749199
- [Background] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941